CLINICAL TRIAL: NCT01790464
Title: Glossopharyngeal Nerve Blockade for Awake Videolaryngoscopy Assisted Endotracheal Intubation in the Morbidly Obese
Brief Title: Glossopharyngeal Nerve Block for Awake Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Albert Moore, Assistant Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 11-201-SDR
Record Dates: First submitted 2013-02-11; First posted 2013-02-13 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Morbid Obesity
Keywords: Glossopharyngeal nerve block; Airway anesthesia; Awake intubation
MeSH Terms: conditions — Obesity, Morbid | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NS gauze (Placebo Comparator): Standard airway anesthesia with 20 ml of aerosolized 2% lidocaine and peritonsillar instillation of gauze soaked in normal saline (Control Group)
  Interventions: Drug: placebo
- Lidocaine gauze (Active Comparator): 20 ml of aerosolized 2% lidocaine and peritonsillar instillation of gauze soaked with 2% lidocaine (Glossopharyngeal Group).
  Interventions: Drug: 2% Lidocaine

INTERVENTIONS:
Drug: 2% Lidocaine — 2% lidocaine and peritonsillar instillation of gauze soaked with 2% lidocaine (Glossopharyngeal Group).
  Arms: Lidocaine gauze
Drug: placebo
  Arms: NS gauze

SUMMARY:
Endotracheal intubation of the morbidly obese is often performed awake. This is performed after topical anesthesia of the patient's pharynx and larynx. There are many techniques used to perform topical anesthesia of the patient's airway, which include aerosolization of local anesthesia, topical application of local anesthesia, and nerve blockade using needles and local anesthesia. Reasons for failure of any awake tracheal intubation technique is excess gagging. The most effective method to adequately anesthetize the airway to decrease the amount of gagging is unknown. The investigators wish to assess if the instillation of local anesthesia soaked gauze next to the peritonsillar pillars will decrease the number of gagging episodes during awake video laryngoscopy assisted tracheal intubation of the morbidly obese.

DETAILED DESCRIPTION:
Research design 1.1 Study design Prospective randomized control trial. 1.2 Patients All morbidly obese patient presenting for bariatric surgery at the Royal Victoria Hospital are eligible.

1.3 Exclusions We will exclude any patient with

* moderate to severe systemic illness, i.e. American Society of Anesthesiologists (ASA) score of 4 or higher
* inability to communicate in English or French
* contraindications to the drugs used in the study 1.4 Recruitment Eligible patients admitted to Royal Victoria Hospital who do not have any of the exclusion criteria will be approached by one of the investigators in the recovery room, or in the preoperative clinic before the scheduled surgery. The study protocol will be explained and a consent form will be given to the patients. Patients will have time and opportunity to ask any questions before the consent will be signed.

1.5 Study protocol Patients will be prepared for surgery according to the routine guidelines established by the Departments of Surgery and Anesthesia at the Royal Victoria Hospital.

They will have an IV and peripheral arterial line inserted, and will have Canadian Anesthesia Society standard monitors placed. Glycopyrrolate 0.4 mg iv will be given to decrease secretions. Using a computer generated randomization table, patients will be assigned to a group that receives standard airway anesthesia with 20 ml of aerosolized 2% lidocaine and peritonsillar instillation of gauze soaked in normal saline (Control Group) or that receives 20 ml of aerosolized 2% lidocaine and peritonsillar instillation of gauze soaked with 2% lidocaine (Glossopharyngeal Group). Sedation will be administered using a remifentanyl intravenous infusion of 0.05 /min with an initial bolus of 0.4µg/kg, and intravenous midazolam 0.05 mg/kg. We will review the chart to obtain patient demographic data including patient age, height, weight, medications, and past medical histories. Baseline blood pressure, heart rate, will be recorded, and a blood sample will be drawn for lidocaine level.

Once the airway is topicalized and sedation has taken effect, the anesthesiologist will insert the video laryngoscope into the patient's oropharynx. Once the ideal view of the vocal cords is obtained, an endotracheal tube fitted with a stylet will be introduced into the pharynx, and then slid through the vocal cords into the trachea. During the intubation attempt, a blinded observer will record the blood pressure and heart rate at every minute, and the best view obtained with the laryngoscope. The observer will assign the patient a reaction score (4) at three time points: the insertion of the video laryngoscope, the pharyngeal insertion of the tracheal tube, and the tracheal insertion of the tracheal tube. This score will be:

1. No reaction
2. Single change in facial expression
3. Grimacing facial expression
4. Severe facial grimace, no reflex head movements
5. Severe facial grimace with head movements
6. Severe facial grimace with head and limb movements The observer will also record the time from the insertion of the video laryngoscope, and the first evidence of endtidal carbon dioxide from the tracheal tube. If the intubation attempt results in a reaction score of 6, or in an inadequate laryngeal view, the treating anesthesiologist may secure the airway in any way they see fit, which may include addition of more topical anesthesia, more sedation, or the use of another airway technique. The number of attempts at intubation, and any other techniques used for intubation will be recorded. We will measure lidocaine levels in blood samples every 10 minutes for 40 minutes after the commencement of the airway anesthesia, using the mass spectrometry method previously used for similar studies at the Royal Victoria Hospital.

ELIGIBILITY:
Inclusion Criteria:

* All morbidly obese patient presenting for bariatric surgery at the Royal Victoria Hospital are eligible.

Exclusion Criteria:

* moderate to severe systemic illness, i.e. American Society of Anesthesiologists (ASA) score of 4 or higher
* inability to communicate in English or French
* contraindications to the drugs used in the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2012-04; Primary Completion 2013-06 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Gag score | 10 minutes
  We wish to assess if the instillation of local anesthesia soaked gauze next to the peritonsillar pillars will decrease the number of gagging episodes during awake video laryngoscopy assisted tracheal intubation of the morbidly obese.

SECONDARY OUTCOMES:
Lidocaine serum level | 40 minutes
  Level of lidocaine in patients serum at 10, 20, 30 and 40 minutes post chewing.